CLINICAL TRIAL: NCT02988089
Title: Efficacy of Two Antimicrobial Susceptibility Testing Guided Antibiotic Selection Strategies in Salvage Helicobacter Pylori Treatment
Brief Title: Antimicrobial Susceptibility Testing Guided Antibiotic Selection Strategies in Salvage Helicobacter Pylori Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); General Hospital of Jinan Military Region (Unknown); Binzhou People's Hospital (Other); Liaocheng People's Hospital (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016SDU-QILU-23
Record Dates: First submitted 2016-12-04; First posted 2016-12-09 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Helicobacter Pylori Infection; Antimicrobial Susceptibility Testing
Keywords: Helicobacter Pylori Infection; Antimicrobial susceptibility testing (AST)
MeSH Terms: interventions — Amoxicillin; Clarithromycin; Metronidazole; Tinidazole; Levofloxacin; Furazolidone; Tetracycline; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- clarithromycin dependant group (Experimental): Patients in this group will receive 14-day bismuth-based quadruple therapies guided by the susceptibility of clarithromycin. Ilaprazole 5 mg b.i.d is used as the proton pump inhibitor (PPI). The dose of colloidal bismuth pectin is 200 mg b.i.d.
  The kinds of 2 antibiotics will be depend on the susceptibility of clarithromycin.
  If clarithromycin is susceptible, amoxicillin 1 g b.i.d and clarithromycin 500 mg b.i.d will be chosen; If clarithromycin is resistant, amoxicillin 1 g bid and furazolidone 100 mg b.i.d will be chosen.
  Interventions: Drug: Clarithromycin susceptibility dependant strategy; Drug: proton pump inhibitor (PPI) and Colloidal Bismuth Pectin; Drug: amoxicillin and clarithromycin or amoxicillin and furazolidone
- 6 antibiotics dependant group (Experimental): Patients in this group will receive a 14-day bismuth-based quadruple regimen to eradicate H. pylori. The regimen is consist of a PPI, a bismuth and 2 susceptible antibiotics which are determined by AST. The susceptibility of amoxicillin, clarithromycin, metronidazole, tinidazole,levofloxacin, furazolidone and tetracycline will be evaluated.
  Ilaprazole 5 mg b.i.d is used as the proton pump inhibitor (PPI). The dose of colloidal bismuth pectin is 200 mg b.i.d.
  Interventions: Drug: 2 susceptible antibiotics (amoxicillin, clarithromycin, metronidazole, tinidazole,levofloxacin, furazolidone and tetracycline ); Drug: proton pump inhibitor (PPI) and Colloidal Bismuth Pectin
- salvage therapy for negative culture (Other): when the results of culture are negative, patients will receive Ilaprazole 5 mg, amoxicillin 1 g, furazolidone 100 mg, Colloidal Bismuth Pectin 200 mg (IAFB regimen) or Ilaprazole 5 mg, amoxicillin 1 g, furazolidone 100 mg, tetracycline 750 mg (IAFT regimen)，all are used twice daily except tetracycline which is taken 3 times daily.
  Interventions: Drug: proton pump inhibitor (PPI) and Colloidal Bismuth Pectin; Drug: amoxicillin and furazolidone or amoxicillin and tetracycline
- salvage therapy for failed eradication (Other): If failed with AST guided eradication therapy, patients will take another therapy according to the former AST results. One susceptible antibiotics not involved in last therapy will be used as a component of 14-day bismuth-based quadruple regimen with Ilaprazole 5 mg b.i.d, amoxicillin 1 g b.i.d and Colloidal Bismuth Pectin 200 mg b.i.d.
  Interventions: Drug: proton pump inhibitor (PPI) and Colloidal Bismuth Pectin; Drug: amoxicillin and furazolidone or amoxicillin and Tinidazole or amoxicillin and Levofloxacin

INTERVENTIONS:
Drug: Clarithromycin susceptibility dependant strategy — Patients in this group will receive a 14-day bismuth-based quadruple regimen to eradicate H. pylori. Antimicrobial susceptibility testing (AST) will be used to test the susceptibility of clarithromycin.
  If clarithromycin is susceptible, amoxicillin 1 g b.i.d and clarithromycin 500 mg b.i.d will be chosen; If clarithromycin is resistant, amoxicillin 1 g bid and furazolidone 100 mg b.i.d will be chosen.
  Arms: clarithromycin dependant group
Drug: 2 susceptible antibiotics (amoxicillin, clarithromycin, metronidazole, tinidazole,levofloxacin, furazolidone and tetracycline ) — Patients in this group will receive a a 14-day bismuth-based quadruple regimen to eradicate H. pylori. The regimen is consist of a PPI, Colloidal Bismuth Pectin and 2 susceptible antibiotics which are determined by AST. The susceptibility of amoxicillin, clarithromycin, metronidazole, tinidazole,levofloxacin, furazolidone and tetracycline will be evaluated.
  Arms: 6 antibiotics dependant group
Drug: proton pump inhibitor (PPI) and Colloidal Bismuth Pectin — all patients need these two drugs.
Drug: amoxicillin and clarithromycin or amoxicillin and furazolidone — patients in the 6 antibiotics dependant group will use these intervention.
  Arms: clarithromycin dependant group
Drug: amoxicillin and furazolidone or amoxicillin and tetracycline — salvage therapy for negative culture when the results of culture are negative
  Arms: salvage therapy for negative culture
Drug: amoxicillin and furazolidone or amoxicillin and Tinidazole or amoxicillin and Levofloxacin — salvage therapy for failed eradication if failed with AST guided eradication therapy
  Arms: salvage therapy for failed eradication

SUMMARY:
Helicobacter pylori (H. pylori), which infects about 50% of the global population, has been recognized as a main risk factor of multiple gastric pathologies, especially non-cardiac gastric cancer. Strongly evidence supports that H. pylori eradication is an effective approach to reduce the incidence of those pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who are 18-70 years old with persistent H. pylori infection after first or second line treatment attempts.

Exclusion Criteria:

* Enable to undergo upper endoscopy;
* Patients with gastrectomy, acute GI bleeding and advanced gastric cancer;
* Known or suspected allergy to study medications;
* Taking bismuth and antibiotics in the previous four weeks, or taking proton pump inhibitor and H2-receptor blockers in the previous two weeks;
* Currently pregnant or lactating
* Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Eradication rates in 2 groups | 6 months

SECONDARY OUTCOMES:
the rate of improving dyspepsia symptoms after H. pylori eradication | 6 months
the rate of adverse events happening | 6 months
the rate of good compliance (take pills more than 90%) | 5 months
difference of cost per patient for each eradication achieved in 2 groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Yanqing, MD, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Ji'nan, Shandong, China

IPD SHARING:
Plan to Share IPD: No